CLINICAL TRIAL: NCT07081399
Title: the Effect of Adult Intubated Patient Clinical Pathway on Post-extubation Complications Prevention
Acronym: CP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Heba.Attia@nur.dmu.edu.eg, assistant lecturer critical care and emergency nursing, Damanhour University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1a2b3c4d5e6f7g8h9i10j11k12l13m
Record Dates: First submitted 2025-01-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Dysphagia; Dysphagia Rehabilitation
Keywords: post-extubation dysphagia; post-extubation laryngospasm
MeSH Terms: conditions — Deglutition Disorders | interventions — Methylprednisolone

STUDY DESIGN:
Intervention Model Description: non- clinical pathway group and clinical pathway group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: post-extubation complications outcomes (laryngospasm, laryngeal edema and dysphagia)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- non-clinical pathway group (No Intervention): non-clinical pathway group who received the routine hospital care.
- clinical pathway group (Experimental): the clinical pathway group who recieved the CP interventions such as: ETTcuff pressure measurement, ETT suctioning, measures to prevent laryngeal edema, swallowing rehabilitation, maneuvers to prevent laryngospasm

INTERVENTIONS:
Combination Product: ETT cuff pressure monitoring, ETT suctioning, cough augmentation technique, swallowing exercises,: Nebulized budesonide 1mg and IV methylprednisolone 40 mg we — cough augmentation, larson maneuver, swallowing rehabilitation

SUMMARY:
Post- extubation complications delay the complete recovery of critically ill patient. The clinical pathway is one strategies that help to manage and control these complications.

DETAILED DESCRIPTION:
The presence of endotracheal tube is associated with various fatal complications which are diagnosed mainly in post- extubation time. Those complications include laryngeal edema, laryngospasm, and post-extubation dysphagia which delay the complete recovery of critically ill patient. The clinical pathway is one of the excellent strategies that help the critical care staff to manage and control these complications

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years)
* orally intubated patients for the first time attached with MV for less than two weeks
* with Glasgow coma scale (GCS) from 13-15.

Exclusion Criteria:

* patients admitted with high risk for laryngeal edema,
* difficult intubation,
* ETT/anterior-posterior diameter ˃45%,
* self-extubation, and
* planned for tracheostomy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
prevention of laryngeal edema | 72 hours after extubation
  measured by respiratory distress observation score that it ranges from 0-16. the high score indicates sever respiratory distress
laryngospasm | 72 hours after extubation
  measured by four point scale. it composed from 4 grades, grade 0 indicates no laryngospasm, grade 3 indicates severe degree of laryngospasm.
dysphagia | 72 hours after extubation
  measured by Gugging Swallowing Screen scale that it ranges from 0 -20. the high score indicates severe dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: sahar youness effect of adult intubated CP on post-extubation complications, Study Chair
Locations (1):
- Faculty of Nursing, Damanhour University, Damanhūr, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No